CLINICAL TRIAL: NCT00582699
Title: Depression, Cytokines and Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); New York Presbyterian Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 05-117; NIH CA102201
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Pancreatic
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (4):
- 1: Patients with pancreatic cancer who meet DSMIV criteria for a current diagnosis of a Major Depressive Episode (N=25).
  Interventions: Behavioral: assessment interview and blood draw
- 2: Patients with pancreatic cancer who do not meet DSMIV criteria for a current diagnosis of Major Depressive Episode (N=25)
  Interventions: Behavioral: assessment interview and blood draw
- 3: Healthy controls who meet DSMIV criteria for a current diagnosis of Major Depressive Episode (N=25).
  Interventions: Behavioral: assessment interview and blood draw
- 4: Healthy controls who do not meet DSMIV criteria for a current diagnosis of Major Depressive Episode (N=25).
  Interventions: Behavioral: assessment interview and blood draw

INTERVENTIONS:
Behavioral: assessment interview and blood draw — All subjects will be administered a battery of clinician rated and self report instruments including measures of depression, fatigue, and cognitive functioning. In addition, measures of pain, sleep, and anxiety will also be utilized to assess these important potential confounding variables. The SCIDIV will be used to ascertain the presence or absence of a current DSMIV diagnosis of Major Depressive Episode for all subjects. The interview should take approximately fortyfive minutes to complete. Patients will have their blood drawn once, in order to determine plasma levels of the cytokines IL1, IL6, TNFalpha, IL10, IL15 and IFNgamma.

SUMMARY:
The purpose of this study is to measure certain specific chemicals in your blood, produced by the body in response to a stress, such as having pancreatic cancer. These chemicals are called "cytokines" and the researchers doing this study want to look at the role they may play in developing depression.

DETAILED DESCRIPTION:
Pancreatic cancer is the 5th leading cause of cancer mortality in the United States, with a 5 year mortality rate of over 95%. With limited treatments available for cure or prolongation of survival, quality of life issues, such as the optimal treatment and understanding of depression, become an important focus of care in this population. Clinical Depression (Major Depressive Syndrome) occurs in up to 50% of patients with pancreatic cancer, and is significantly more common than in other cancers. Accumulating evidence suggests a potential role for endogenous cytokines, specifically interleukin-1 (IL-1), interleukin-6 (IL-6) and tumor necrosis factor alpha (TNF-alpha) in the development of depression in the medically ill, including cancer patients. These same cytokines have been noted to be elevated in pancreas cancer patients. The main goal of this pilot study is to examine the role of specific endogenous cytokines (IL-1, IL-6, TNF-alpha, as well as IL-10, Il-15 and IFN-gamma) in the development of Major Depressive Syndrome (MDS) in patients with pancreatic cancer. To achieve our goal, we will examine the relationships between serum cytokines (IL-1, IL-6, TNF-alpha, as well as IL-10, Il-15 and IFN-gamma) and clinical depression (i.e. MDS) utilizing a cross sectional design in 4 samples of patients: a) Pancreas cancer patients with a DSM-IV diagnosis of MDS (N=25); b) Pancreas cancer patients without a DSM-IV diagnosis of MDS (N=25); c) Healthy Controls with a DSM-IV diagnosis of MDS (N=25); and d) Healthy Controls without a DSM-IV diagnosis of MDS (N=25). Measures will include a structural clinical interview for DSM-IV diagnosis (SCID) of Major Depressive Syndrome, as well as measures of depressive symptom severity, fatigue severity, concentration and attention, and cognitive function. Plasma concentrations of endogenous cytokines ((IL-1, IL-6, TNF-alpha, as well as IL-10, Il-15 and IFN-gamma) will be measured utilizing standard assays. Our specific aims are: 1) To preliminarily examine the relationships between plasma concentrations of endogenous cytokines (IL-1, Il-6, TNF-alpha, as well as IL-10, Il-15 and IFNgamma) and a DSM-IV diagnosis of Major Depressive Syndrome in patients with pancreas cancer and healthy controls; 2) To explore the relationships between plasma concentrations of endogenous cytokines (Il-1, Il-6, TNF-alpha, as well as IL-10, Il-15 and IFN-gamma) and the phenomenology and severity of depressive symptoms, presence and severity of fatigue, and degree of impairment in attention, concentration and cognition, in depressed patients with pancreas cancer and healthy depressed controls. The results of this pilot study will be utilized to seek NIH funding for larger, longitudinal, multi-institutional, studies examining the role of endogenous cytokines in pancreas cancer patients, as well as clinical intervention trials for the treatment of clinical depression in pancreas cancer patients that utilize specific cytokine antagonists as adjuncts to antidepressant drug therapies.

ELIGIBILITY:
Inclusion Criteria:

1. 40 years of age or older at the time of recruitment.
2. Unresectable/inoperable pancreatic adenocarcinoma (stage III or IV), receiving Gemcitabine or Gemcitabine-based combination therapy.
3. If in the "depressed" sample, patients with pancreatic cancer must meet DSM-IV criteria for a major depressive syndrome (based on the SCID) AND have an HDRS score of 18 or greater.
4. If in the "non-depressed" sample, patients with pancreatic cancer must not meet DSM-IV criteria for a major depressive syndrome (based on the SCID) AND must have a HDRS score of 17 or less.

Exclusion Criteria:

1. A. Patient has reported experiencing or medical record indicates a serious medical event (i.e.,medical hospitalization (excluding hospitalization related to cancer diagnosis/treatment),myocardial infarction, stroke) within the year preceding study participation.

B. Patient has reported the presence of or medical record indicates:

* Type 1 Diabetes, unrelated to cancer diagnosis
* renal failure requiring dialysis
* inflammatory bowel disease 3. Patient has reported the presence of or medical record indicates an active secondary cancer diagnosis, however patients who have been treated for a past cancer and are 2 years disease free from that cancer can participate.

  4. Presence of a medical/surgical condition obtained through self-report associated with elevated cytokine levels, such as:
* HIV/AIDS
* Auto-immune diseases such as SLE, Multiple Sclerosis, Rheumatoid Arthritis, Polymyalgia Rheumatica, Temporal Arteritis, Chronic Fatigue Syndrome, severe allergies
* Congestive Heart Failure
* Recent stroke
* Alzheimer's Disease
* Active infection;
* Acute pancreatitis
* Acute pericarditis
* Acute hepatitis including Hepatitis C
* Recent vaccination for viral disease
* Major surgery within the past 6 weeks

  5. Patient Reports Receiving treatment (within two weeks) with:
* Interleukin
* Interferon
* Thalidomide
* NSAID's
* Cox-2 inhibitors
* Cancer vaccine therapies

  6. Self-reported diagnosis with a major psychiatric disorder other than depression (e.g. psychosis secondary to Bipolar Disorder, Schizophrenia, Schizo-affective illness, substance abuse) so severe that, in the opinion of the study staff, would interfere with a patient's ability to give informed consent for research.

  7. Cognitive impairment so severe that, in the opinion of the study staff, would interfere with a patient's ability to give informed consent or complete study measures for research.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruitment of patients will take place primarily in the Ambulatory Care Facility on 53rd street in the GI Oncology Clinic treating pancreatic cancer.
  Healthy control subjects with depression will be recruited from the New York Hospital Payne Whitney Clinic outpatient facilities and MSKCC. Healthy control subjects without depression will be recruited from contacts supplied by study participants (e.g. spouses, relatives and friends) and from Memorial Hospital staff volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2005-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The levels of specific cytokines (IL-1, Il-6, TNF-alpha, as well as IL-10, Il-15 and IFN-gamma), the diagnosis of Depression, depressive symptom severity, and the pattern of depressive symptoms. | November 2010

CONTACTS AND LOCATIONS:
Overall Officials: Williams Breitbart, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center website — http://www.mskcc.org